CLINICAL TRIAL: NCT03044483
Title: Establishing Normal Ranges of Microcirculatory Function as Determined by CytoCam-IDF Imaging
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 214674
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Microcirculation
Keywords: Sepsis; Microcirculatory function
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 18-34 year olds: Healthy adults aged 18-34 years old
  Interventions: Other: Measurement of sublingual microcirculatory parameters
- 35-54 year olds: Healthy adults aged 35-54 years old
  Interventions: Other: Measurement of sublingual microcirculatory parameters
- 55 and over year olds: Healthy adults aged 55 years old and over
  Interventions: Other: Measurement of sublingual microcirculatory parameters

INTERVENTIONS:
Other: Measurement of sublingual microcirculatory parameters — Measurement of the sublingual microcirculatory function using the CytoCam-IDF imaging device to establish the normal range for each age group noted.

SUMMARY:
When infection strikes, the body's immune system reacts by producing chemicals in the bloodstream and changes in white blood cells to attack the infecting organism (bacteria, viruses or other organisms) and prevent it spreading. This is termed the 'inflammatory response'. Though beneficial in fighting infection, this response can sometimes be excessive, causing harmful effects on body organs. This is termed the 'systemic inflammatory response syndrome' and when linked to infection is termed 'sepsis'.

Previous research has shown that in patients who have sepsis, the small blood vessels supplying oxygen and nutrients to muscles and other organs (the microcirculation) become abnormal and do not function as they would in health. However, it is difficult to assess the function of microcirculation in clinical practice, and we want to find new, easier ways of doing so.

The aim of this study is to test a new method for assessing the function of these small blood vessels, by directly visualising them using a highly sensitive microscope, the size of a pen, placed under the tongue. By understanding the flow of blood in these vessels in healthy individuals, we will gain a better understanding of how these vessels are affected in illness.

DETAILED DESCRIPTION:
Background

Sepsis is a highly heterogeneous disease state brought about by a dysregulated host response to systemic infection, with uncontrolled pro- and anti-inflammatory processes leading to collateral tissue injury and immune suppression.

Sepsis poses a significant health burden worldwide, with deaths attributed in the UK estimated at approximately 44,000 per annum. Prompt treatment directed by internationally agreed management guidelines improves outcomes in sepsis. However early diagnosis of sepsis remains difficult, with current diagnostic criteria relying on the presence of organ dysfunction and derangement of macro haemodynamic variables. At the point of diagnosis, mortality is in excess of 10%. At present there are no specific criteria in the diagnosis of sepsis based on the underlying pathophysiological abnormalities, specifically on assessment of the microcirculation.

The microcirculation in sepsis

The microcirculation consists of a dense network of arterioles, capillaries and venules, whose diameter is less than 150 um. Its functions are to supply nutrients and oxygen for aerobic metabolism and to reduce cellular waste products.

Sepsis affects all elements of the microcirculation, with microcirculatory dysfunction playing an important role in the pathophysiology of severe sepsis and septic shock. Sepsis is associated with decreased capillary density and increased perfusion heterogeneity leading to decreased oxygen delivery, tissue hypoxia and subsequently organ dysfunction. Changes in microcirculatory function may precede the traditional diagnostic features of sepsis, providing earlier information on patients who will go on to develop severe sepsis and multi-organ failure. Recognition of sepsis at this early stage would allow prompt treatment, aimed at restoring homeostasis of the microcirculation, therefore altering disease progression.

A number of studies have demonstrated that improvements in microcirculatory function following early resuscitation are associated with decreasing organ dysfunction, and those patients whose microcirculations fails to improve following resuscitation have poorer outcomes. Despite recognition of the importance of the microcirculation in sepsis, current goal-directed end points rely on the monitoring and restoration of global measures of cardiovascular/organ function (e.g. heart rate, blood pressure, urine output, lactate), partly because the microcirculation is difficult to monitor in clinical practice. However, improvement in macro haemodynamic variables does not guarantee restoration of microcirculatory homeostasis. Clinical assessment of microcirculatory function is presently inferred from the measurement of by-products generated due to impaired oxygenation/metabolism such as lactate and carbon dioxide.

Video microscopic techniques for assessment of the microcirculation

Video microscopic techniques provide in-vivo visualisation of the microcirculation, allowing direct measurement of capillary density, perfusion and flow dynamics. Until recently, these techniques which have included Orthogonal Polarization Spectral (OPS) imaging and Sidestream Dark Field (SDF) imaging, have been clinically inaccessible owing to their bulky nature, operator dependant output and time-consuming offline analysis requirement.

A third-generation handheld microscope has recently been developed (CytoCam-IDF, Braedius Medical, NL), utilising Incident Dark Field (IDF) illumination. The device incorporates real-time automated digital image analysis, combined with high resolution lenses and a computer controlled image sensor for improved resolution. The CytoCam also features a novel quantitative focusing mechanism with an integrated distance measuring system, whereby once the focus depth has been established for a specific patient, serial measurements can be made without having to manually readjust the focus, improving speed and ease of measurements. This new device performs well when compared to previous devices, providing improved contrast and image sharpness allowing an increased number of microvessels to be visualised.

Crucially, the CytoCam is equipped with bespoke software allowing images to be stored and analysed automatically at the point of acquisition. Microcirculatory monitoring is a not a new technique, but the combination of user friendly ergonomics, accurate image acquisition and automated analysis opens up this potentially useful direct measurement of microcirculatory function to bedside clinical practice.

Analysis of the sublingual microcirculation A round table discussion in 2006 by experts in the field, sought to clarify the features that should be included in microcirculatory analysis, concluding that assessment of the microcirculation should include measures of vascular density, assessment of capillary perfusion and a heterogeneity index (in vessels of <20 micrometres in diameter).

These measured variables are:

Microvascular Flow Index (MFI) - Perfusion quality Image divided in to quadrants. A number is assigned to each quadrant according to predominant flow type (0 = no flow, 1 = intermittent, 2 = sluggish, 3 = continuous). The MFI results from the mean of the 4 values.

Total Vessel Density (TVD) Vessel density - The total length of the vessels divided by the total surface area of the analysed area.

Perfused Vessel Density (PVD) - Functional vessel density Total length of perfused vessels (MFI score 2/3) divided by the analysed area.

Proportional of Perfused Vessels (PPV) - Perfusion quality 100 x number of perfused vessels divided by the total number of vessels Heterogeneity Index (HI) Measure of the heterogeneity of flow between vessels. Highest MFI - lowest MFI divided by mean MFI across all sites analysed

Compared to healthy volunteers, patients with sepsis display lower values for PVD, PPV and MFI, along with increased heterogeneity index, irrespective of macro haemodynamic condition. Total capillary density appears to be unaffected by sepsis. These findings were corroborated by the International Study on Microcirculatory Shock Occurrence in Acutely Ill Patients (microSOAP) study.

The microSOAP study is to date the largest trial investigating the significance of microcirculatory alterations in a heterogeneous ICU population (i.e. not just those with sepsis). Using the previous generation of similar technology, the investigators found that of the 501 patients included for analysis, 86 (17%) had an abnormal MFI (defined a priori as <2.6). Of those with an abnormal MFI, the HI was increased with decreased PPV and PVD. Total vessel density was not affected. Abnormal MFI in conjunction with tachycardia was associated with an increased mortality (OR 3.24).

CytoCam Tools automated analysis

CytoCam Tools is the proprietary software supplied with the aforementioned microcirculatory monitor. It utilises a new analysis technique termed Capillary Network Analysis (CNA) whereby the microcirculation is analysed automatically and in a user-independent nature by a two-stage process which includes automatic vessel detection (depending on the diameter of visualised vessels), followed by an assessment of speed of red blood cells in the vessels identified.

The following microcirculatory variables are then automatically determined.

* Total Vessel Density (TVD) - Total length of all detected vessels divided by the processed area.
* Speed Index (SI) - Relative number derived from the intensity variation along the centreline of a vessel, which describes the speed detected in the vessel.
* Perfused Speed Index (PSI) - SI in a vessel where the SI is higher than the perfusion threshold (PT).
* Average Perfused Speed Indicator (APSI) - Sum of all PSI values divided by the total number of perfused vessels.
* Proportion of perfused vessels (PPV) - Total length of all vessels with an SI higher than the PT, divided by the total length of all detected vessels x 100,
* Perfused Vessel Density (PVD) - Total length of all vessels with an SI higher than the PT divided by the processed area.
* Average Perfused Speed Indicator Heterogeneity Index (APSI HI) - Image divided in to quadrants and APSI derived for each quadrant. APSI highest minus the lowest APSI divided by the mean APSI of all quadrants.

The assessment of PPV and PVD relies on the automated analysis of red blood cell speed in identified vessels. In order to achieve this a predetermined Perfusion Threshold (PT) is set. The PT describes the state of flow within identified vessels and can range from 0 to infinite. Manufacture assessment has determined that a PT of over 1 is consistent with a "perfused condition" and this can be subdivided further as follows:

Perfusion threshold

State of flow 0 - 1 = No flow 1 - 5 = Sluggish 5 or greater = Good flow Normal ranges for these automatically measured variables in health are currently unknown. Understanding the normal ranges would allow us to utilise this technique in future studies concerning the early diagnosis of septic illness. Identification of patients at an early stage in the pathophysiological process of sepsis before the development of traditionally diagnostic macro-circulatory abnormalities may allow earlier implementation of treatment.

Rationale

The CytoCam system may represent a step towards a more user-friendly, reproducible, clinically applicable approach to measuring, and acting upon changes in microvascular function to improve clinical outcomes. However, the normal ranges for these measurements are not known, without which further studies cannot take place. This study will identify the normal ranges for the automatically determined measurements derived by the CytoCam system in healthy subjects, and open new opportunities for studies, which we anticipate will be aimed at the early identification of patients with microcirculatory dysfunction (as is found in sepsis); whose microcirculatory parameters fall outside of these newly defined ranges. This will be the first step in moving towards routine bedside microcirculatory monitoring in our intensive care unit.

This work builds on projects currently in progress within the Diagnostic Development Unit (DDU) based at Leicester Royal Infirmary. The DDU is a University of Leicester inter-collegiate project between Medicine, Space Science and Atmospheric Chemistry, exploring the use of novel non-invasive monitors in Emergency Medicine and Critical Care.

Population to be studied

OBJECTIVE

To identify the normal ranges for automatically measured microcirculatory variables as determined by the CytoCam system in different adult age groups.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* No current acute illness
* No changes to chronic medications in the 4-weeks preceding recruitment.
* Able and willing to comply with all study requirements.

Exclusion Criteria:

* Participant aged under 18 years old.
* Participant has an acute illness, as identified by clinical history
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants awaiting maxillofacial surgery for any reason.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults aged 18 years and over, with no acute illness
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Microvascular Flow Index (MFI, No units) | 6 months
  Measurement of MFI in the the three stated age groups
Total Vessel Density (TVD, mm/mm2) | 6 months
  Measurement of TVD in the three stated age groups
Perfused Vessel Density (PVD, mm/mm2) | 6 months
  Measurement of PVD in the three stated age groups
Proportion of Perfused Vessels (PPV, no units | 6 months
  Measurement of PPV in the three stated age groups

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Thompson, MBChB, Principal Investigator — Principal Investigator
Locations (1):
- University Hospitals of Leicester, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No